CLINICAL TRIAL: NCT05470686
Title: Study of the Relationship Between the Relative Variation of PaO2/FiO2 and the Variation of Lung Ultrasound Score During the First Session of Physiotherapy Associated With Non-invasive Ventilation in Cardiac Surgery Patients by Cardiopulmonary Bypass
Brief Title: Study of the Relationship Between the Oxygenation State and Lung Ultrasound Score in Cardiac Surgery
Acronym: PaFiKinESAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Aurelie OUDIN-ROTH, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A01478-35
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Heart Surgery
Keywords: heart surgery; Lung ultrasound score; PaO2/FiO2 ration; physiotherapy; Non invasive ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEART SURGERY PATIENTS with cardio pulmonary bypass (Other)
  Interventions: Biological: blood gas via arterial catheter

INTERVENTIONS:
Biological: blood gas via arterial catheter — Patients will have a blood sample plus a lung ultrasound before and after the physical therapy session combined with non invasive ventilation the morning after the heart surgery
  Other Names: Lung ultrasound score

SUMMARY:
After conventional cardiac surgery, many respiratory complications are possible. Therefore, the resuscitator prescribe physiotherapy and non invasive ventilation. The physiotherapist has few reliable tools to evaluate and follow the patient on his ventilatory function. Currently, lung ultrasound is little used in physiotherapy and no study explains the link between the lung ultrasound results and oxygenation patient state. Before considering the interest of lung ultrasound score as a criterion of effectiveness of a physiotherapy treatment through future studies, it is first important to objectivize the existence of a relationship between lung ultrasound score and the PaO2/FiO2 ratio after cardiac surgery. Lung ultrasound could provide direct clinical information without having to resort to other more invasive examinations to objectify the improvement of the patient's oxygenation.

Main objective To show that the relative change in the PaO2/FiO2 ratio correlates with the change in lung ultrasound score measured in the short term between the beginning and the end of the first physiotherapy session associated with non invasive ventilation the day after surgery in cardiac patients

Secondary objectives

* To study the inter-operator (2 readers) reproducibility of the lung ultrasound score measurement.
* To study the relationship between the relative variation of the PaO2/FiO2 ratio and the variation of each of the 12 zones of the lung ultrasound score
* To Study the relationship between the initial lung ultrasound score and the relative variation of the PaO2/FiO2 ratio
* To study the relative variation of the PaCO2 and the variation of the lung ultrasound score between the beginning and the end of the first session of physiotherapy management associated with NIV
* To obtain from the patient in the short term feedback on his or her understanding of the explanations about lung ultrasound score provided by the physiotherapist during the session

ELIGIBILITY:
Inclusion Criteria:

* Person having received complete information on the organization of the research and having given written consent to participate
* Person having benefited from a heart surgery under cardio-pulmonary bypass
* Medical prescriptions for non invasive ventilation and physiotherapist
* Age ≥ 18 years
* 18.5 ≤ BMI ≤ 35 kg/m2
* Visual Analogy Scale pain < 4
* Patient conscious and oriented: Glasgow 15/15

Exclusion Criteria:

* At the patient's request : a patient may withdraw from the research at any time without affecting the quality of care to which he or she is entitled (withdrawal of consent).
* Cardiorespiratory arrest during the inclusion visit.
* Need for orotracheal reintubation during the inclusion visit.
* Patient non-cooperation during the inclusion visit.
* Failure of the ultrasound machine during the inclusion visit.
* Failure of the blood gas analyzer.
* Glasgow < 15 during the inclusion visit
* PEEP > 6 cmH2O required during physiotherapy + non invasive ventilation session
* PEEP < 6 cmH2O required during physiotherapy + non invasive ventilation session
* Premature interruption of the physiotherapy session + non invasive ventilation not hemodynamically tolerated
* Need for a session of non invasive ventilation + physiotherapy > 30 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Relative difference in PaO2/FiO2 ratio: (measurement after - measurement before the physiotherapy session + non invasive ventilation) / measurement before.) | the morning after the heart surgery
  The higher the ratio, better is the result. Between approximately 0 and 400
Difference in lung ultrasound score: measurement after - measurement before the physiotherapy session + non invasive ventilation | the morning after the heart surgery
  Lung ultrasound score = global measurement on 12 thoracic regions (6 per hemithorax: 2 anteriors, 2 laterals, 2 posteriors) to obtain a result out of 36 (sum of all values found in each zone). Each zone is evaluated as follows:
  0 = normal ventilation
  1. = multiple B-lines defined
  2. = coalescing B-lines
  3. = pulmonary consolidation

SECONDARY OUTCOMES:
Lung ultrasound score values obtained by both evaluators from the same recorded ultrasound images. If there is a difference of one point between the two scores measured, a third reading by a doctor will be taken. This 3rd score will then be retained. | in the week following the measurements
  If there is a difference of one point between the two scores measured, a third reading by a doctor will be taken. This 3rd score will then be retained.
relative difference in PaO2/FiO2 ratio | the morning after the heart surgery
  The higher the ratio, better is the result. Between approximately 0 and 400
difference in lung ultrasound score for each study area | the morning after the heart surgery
  Each zone is rated from 0 to 3 points. The lower the score, the better the result. We look to see if the score for each zone decreases between before and after the physiotherapy session.
initial lung ultrasound score | the morning after the heart surgery
  Lung ultrasound score = global measurement on 12 thoracic regions (6 per hemithorax: 2 anteriors, 2 laterals, 2 posteriors) to obtain a result out of 36 (sum of all values found in each zone). Each zone is evaluated as follows:
  0 = normal ventilation
  1. = multiple B-lines defined
  2. = coalescing B-lines
  3. = pulmonary consolidation
relative difference in PaCO2 | the morning after the heart surgery and after physiotherapy session
  The lower the score, the better the result. Ap proximately between 0 and 100
For each subject, answers to two questions at the end of the session about his or her understanding of PAS after the information provided by the MK during the session | the morning after the heart surgery
  Questions asked by the physiotherapist for the patient (at the end of the session) :
  1. Did you understand the explanations provided by the physiotherapist regarding the lung ultrasound results? Yes, completely Yes, partially No No answer
  2. Did the explanations provided by the physiotherapist regarding the results of the lung ultrasound score help you understand the movements or displacements that the physiotherapist asked you to make during this session? Yes, completely Yes, partially No No answer
  Translated with www.DeepL.com/Translator (free version)

CONTACTS AND LOCATIONS:
Overall Officials: Jean PAYSANT, Study Director — Central Hospital, Nancy, France
Locations (1):
- centralHNF, Vandœuvre-lès-Nancy, France